CLINICAL TRIAL: NCT02906228
Title: Einfluss Hochfrequenter Elektromagnetischer Felder Auf Gehirnaktivität, Schlaf Und Kognitive Leistungsfähigkeit älterer Frauen
Brief Title: Radiofrequency Electromagnetic Field (RF-EMF) Effects on Brain Activity During Sleep and Waking in Healthy Elderly Women
Acronym: EMF60+women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Federal Office for Radiation Protection, Germany (Other Government)
Collaborators: Seibersdorf Labor GmbH (Industry)
Responsible Party: Principal Investigator, Heidi Danker-Hopfe, Ph.D., Head of Competence Center of Sleep Medicine, The Federal Office for Radiation Protection, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3614S30012
Record Dates: First submitted 2016-08-24; First posted 2016-09-20 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Nervous System Effects
Keywords: non-ionizing radiation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSM 900 MHz (Experimental): Radiation: Exposure within the given regulatory limits for non-ionizing electromagnetic fields according to ICNIRP guidelines and German law
  Interventions: Radiation: Exposure within the given regulatory limits for non-ionizing electromagnetic fields according to ICNIRP guidelines and German law
- TETRA 385 MHz (Experimental): Radiation: Exposure within the given regulatory limits for non-ionizing electromagnetic fields according to ICNIRP guidelines and German law
  Interventions: Radiation: Exposure within the given regulatory limits for non-ionizing electromagnetic fields according to ICNIRP guidelines and German law
- Sham Exposure (Experimental): Radiation: Exposure within the given regulatory limits for non-ionizing electromagnetic fields according to ICNIRP guidelines and German law
  Interventions: Radiation: Exposure within the given regulatory limits for non-ionizing electromagnetic fields according to ICNIRP guidelines and German law

INTERVENTIONS:
Radiation: Exposure within the given regulatory limits for non-ionizing electromagnetic fields according to ICNIRP guidelines and German law

SUMMARY:
The purpose of this study is to investigate possible effects of radio frequency electromagnetic fields on EEG activity during sleep and on Brain function during wake (EEG in the resting state condition, slow EEG potentials, auditory evoked potentials) and cognitive performance measures in test of selective attention, divided attention and working memory in healthy elderly females (60 - 80 years).

DETAILED DESCRIPTION:
To investigate possible effects of radio frequency electromagnetic fields on EEG activity during sleep and on Brain function during wake (EEG in the resting state condition, slow EEG potentials, auditory evoked potentials) and cognitive performance measures in test of selective attention, divided attention and working memory in healthy elderly females (60 - 80 years).

Subjects will be exposed with signals from mobile communication handheld devices for 7.5 h during the night and for the whole duration of the test session during the day. Exposures will be GSM (900 MHz), TETRA (400 MHz) and sham. Each subject is exposed with each exposure three times in addition to an adaptation/screening night and day to learn the test.

The results have to be discussed in the context of possible health risks resulting from RF

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects (age 60 - 80 years) right handedness alpha EEG as resting state EEG

Exclusion Criteria:

* acute illness severe neurological, psychiatric or internal disease CNS active medication sleep disorders drug abuse

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04-01; Primary Completion 2016-12-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
sleep assessed by EEG power | during 8 h exposure

SECONDARY OUTCOMES:
restin g state waking EEG (Power) | during exposure 4 h

CONTACTS AND LOCATIONS:
Overall Officials: Blanka Pophof, Ph.D., Study Director — Federal Office of Radiation Protection
Locations (1):
- Competence Center Sleep Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danker-Hopfe H, Dorn H, Sauter C, Schmid G, Eggert T. An experimental study on effects of radiofrequency electromagnetic fields on sleep in healthy elderly males and females: Gender matters! Environ Res. 2020 Apr;183:109181. doi: 10.1016/j.envres.2020.109181. Epub 2020 Jan 24. PMID 32014649